CLINICAL TRIAL: NCT04254757
Title: Percutaneous Endoscopic Decompression for Lumbar Canal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Xuanwu Hospital, Beijing (Other); Beijing Changping Hospital (Unknown)
Responsible Party: Principal Investigator, Liu xiaoguang, PH.D.,M.D.,Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BYSYZD2019001
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Spinal Stenosis; Surgery
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous endoscopic surgery group (Other)
  Interventions: Procedure: Two different treatment
- Open decompression and fusion surgery group (Other)
  Interventions: Procedure: Two different treatment

INTERVENTIONS:
Procedure: Two different treatment — One group treated by percutaneous endoscopic surgery. The another group treated by open decompression and fusion surgery

SUMMARY:
Lumbar spinal stenosis (LSS) is the most common spinal degenerative disease. For conservative treatment failure, open lumbar decompression and fusion surgery is the main surgical treatment. After decades of development, open lumbar decompression and fusion surgery has been the standard treatment. However, there are still people and conditions that cannot be covered, such as elderly people who intolerable surgery, severe osteoporosis, and re-stenosis at adjacent segments after fusion. Percutaneous spinal endoscopic lumbar spinal decompression technique could be performed under local anesthesia, soft tissue damage is minimized, and effective spinal decompression can be achieved. There are still some controversial points of LSS decompression under percutaneous endoscope surgery, such as the range of decompression, choice of approach, postoperative spinal stability, learning curve, surgical safety, long-term effects of endoscopic treatment of restenosis at adjacent segments after fusion surgery. The purpose of this study was to solve these controversial points. A multi-center, prospective registration study based on the real world is planned. The total sample size is about 600 cases (300 cases in endoscopic surgery group, 300 cases in open decompression and fusion group). The mid- to long-term clinical efficacy and safety were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic lumbar canal stenosis(including central canal, lateral recess, foraminal and extraforaminal) despite more than 6 weeks of conservative treatment; Pathology was confirmed by both computed tomography and magnetic resonance imaging The operative level≤2

Exclusion Criteria:

* Segmental instability Simple disc herniation Coexisting pathological conditions, such as tumor and infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified MacNab criteria | 1 years after surgery
Visual Analog Scale (VAS) | at 1 years after surgery
  VAS of leg and back
Oswestry Disability Index(ODI) | at 1 years after surgery

SECONDARY OUTCOMES:
Range of motion(ROM) | at 1 years after surgery
  ROM of operated level
Adjacent Segment Disease | at 1 years after surgery
  Measured on CT and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoguang Liu, M.D.,Ph.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhai S, Zhao W, Zhu B, Huang X, Liang C, Hai B, Ding L, Zhu H, Wang X, Wei F, Chu H, Liu X. The effectiveness of percutaneous endoscopic decompression compared with open decompression and fusion for lumbar spinal stenosis: protocol for a multicenter, prospective, cohort study. BMC Musculoskelet Disord. 2022 May 27;23(1):502. doi: 10.1186/s12891-022-05440-4. PMID 35624443